CLINICAL TRIAL: NCT03771547
Title: ERCP in Super-aged Patients Considering Difficult Cannulation: Challenges and Adverse Events
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: DC-0918
Record Dates: First submitted 2018-10-07; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-02

CONDITIONS: Post-ERCP Acute Pancreatitis; Cholangitis
Keywords: ERCP; Elderly; Difficult cannulation
MeSH Terms: conditions — Cholangitis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- More 80: The first group included ERCP patients aged 80 and above.
  Interventions: Diagnostic Test: ERCP
- Less 80: The second group included those ERCP patients younger than 80.
  Interventions: Diagnostic Test: ERCP

INTERVENTIONS:
Diagnostic Test: ERCP

SUMMARY:
Today 11 percent of China's population is over the age of 65, and according to United Nations, it will take China just 20 years for the proportion of the elderly population to double to 25%. As life expectancy has increased, application of Endoscopic Retrograde Cholangiopancreatography (ERCP) in super-aged (≥80 years of age) is no longer limited with increasing prevalence of choledocholithiasis, and malignancy in advancing age. This increasing may come with more difficulty in cannulation or more complications in senior patients. Regarding difficult cannulation, little is known about grading difficulty in the elderly and its relation with adverse events. Therefore, it is time to evaluate the risk factors of adverse events in super-aged patients with difficult bile duct cannulation.

DETAILED DESCRIPTION:
AIM: To evaluate the incidence, causes, and management of difficult biliary cannulation during ERCP in elderly patients and its role as a risk factor for adverse events.

METHODS: A total of 614 patients, with a mean age of 65.3±16.7 years, underwent ERCP during the study period, were prospectively managed and divided into two groups based on their age. There were 146 patients aged 80 years or older in group A with the mean age of 84±3.4 years. The primary outcome measurements were the difficulty grade of papilla cannulation, clinical outcomes, and ERCP-related complications in the two groups. The adverse events were analyzed by logistic regression about patient age, co-morbidities, indications, and difficult cannulation grading.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent ERCP between July 2016 and January 2018.

Exclusion Criteria:

* We excluded the patients who underwent ERCP for the objectives of follow up, stent removing or taking a biopsy.

Ages: 16 Years to 94 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: No specific restrictions on selecting the patients.
Sampling Method: Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Adverse events in difficult cannulation patients | 30 days
  Multi-variate regression will be used to check the risk factors of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lin Miao, PhD, Principal Investigator — Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tabak F, Ji GZ, Miao L. Impact of periampullary diverticulum on biliary cannulation and ERCP outcomes: a single-center experience. Surg Endosc. 2021 Nov;35(11):5953-5961. doi: 10.1007/s00464-020-08080-8. Epub 2020 Oct 7. PMID 33029732